CLINICAL TRIAL: NCT05266729
Title: A Single Center, Randomized, Placebo Controlled Phase Ⅱ Study to Determine the Dosing Interval and the Optimal Dose of AYP-101 S.C. Injection for the Reduction of Submental Fat
Brief Title: Determine the Dosing Interval and Optimal Dose of AYP-101 for the Reduction of Submental Fat in Chin Area
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AMIpharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AYP-101-202
Record Dates: First submitted 2022-02-15; First posted 2022-03-04 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AYP-101 1 (Experimental): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments.
  Interventions: Drug: Polyene Phosphatidylcholine
- AYP-101 2 (Experimental): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments.
  Interventions: Drug: Polyene Phosphatidylcholine
- Placebo (Placebo Comparator): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Polyene Phosphatidylcholine — Formulated as an injectable solution containing Polyene Phosphatidylcholine at two concentration of 25 mg/mL and 50 mg/mL.
  Other Names: AYP-101
  Arms: AYP-101 1; AYP-101 2
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo

SUMMARY:
To determine the dosing interval, optimal dose, evaluate safety, and efficacy of AYP-101 S.C injection for the reduction of Submental Fat (SMF).

DETAILED DESCRIPTION:
This study is to determine the dosing interval, optimal dose, evaluate safety and efficacy of AYP-101 S.C injection for the reduction of SMF who wish improvement in the appearance of moderate to severe convexity or fullness associated with SMF in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 19 and under 65 years old
* Localized submental fat under chin area and who meet all the following criteria.

  ① Determined as grade 2 (moderate) or 3 (severe) on both using the CR-SMFRS and PR-SMFRS at visit 1

  ② Determined as grade 2 (less satisfied) or less by oneself, using the SSRS at visit 1
* Stable weight over the last 6 months (body weight change within +/-10%), subject who should refrain from exercise and diet that may affect the study results, and who agreed to remain it for the study period
* Singed informed consent

Exclusion Criteria:

* Allergic to beans, components of the clinical drug, or medical devices which used in this clinical trial (lidocaine, acetaminophen, sterile oil pan, alcohol swab, grid pad, needle, etc.)
* Central, endocrine, or hereditary obesity (BMI 35kg/m2 or more)
* History of any treatment (orthognathic surgery, suction lipectomy, PPC or DCA injection) in the neck or chin area
* History of any treatment such as mesotherapy, carboxy, laser surgery, acupuncture needle, filler, chemical peeling with in 1 year, and a botox surgery within 6 months before screening
* Judged to be unsuitable subject for the clinical trials; ① Abnormal or sagging skin, ② Noticeable platysma band under the chin area, ③ Less or short chin than normal ④ Chin or neck disease that are considered to have an impact on the clinical trial such as lymphadenopathy, Inflammation, scars, or surgery on the injection area
* History of or present symptoms of dysphagia
* Heart disease (cardiac insufficiency, angina, cardiac infarction) or stroke within 6 months before screening
* Requiring treatment of joint inflammation or a lung disease
* Uncontrolled hypertension (systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg) or type 2 diabetes mellitus (HbA1c> 9%)
* Type 1 diabetes mellitus who needs insulin treatment
* Autoimmune disorder as well as those who takes immunodepressant drugs
* Hemostatic disorder or those who takes anticoagulant drug such as warfarin and clopidogrel
* Thyromegaly, thyrotoxicosis, or HIV-positive
* Diagnosed with malignant tumor within the last 5 years
* Severe renal dysfunction (serum creatinine > 2.0 mg/dl) or severe dyshepatia (ALT, AST, alkaline phosphatase > maximum rate of normality x 2.5)
* History of serious psychiatric disease (Depression, schizophrenia, epilepsy, alcoholism, drug addiction, anorexia, anorexia nervosa, etc.)
* History of taken a drug that can affect body weight or lipid metabolism such as anorectic agent, steroids, thyroid hormones, amphetamine, cyproheptadine, phenothiazine, or drugs that affect absorption, metabolism, and excretion within 3 months before screening
* History of other clinical trial studies within 6 months before screening
* Women who are pregnant, breastfeeding, having pregnancy plan, or did not agreed to the contraception (contraceptive pills, contraceptive hormones, IUCD, spermicide, condoms etc.)
* Judged to be unsuitable subject for the clinical trials

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who improved at least 1 grade in both Evaluator-Reported Submental Fat Rating Scale (ER-SMFRS) and Subject-Reported Submental Fat Rating Scale (PR-SMFRS) | 4 weeks after the final treatment
  Submental Fat Rating Scale is scored on a 5-point scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.

SECONDARY OUTCOMES:
Percentage of subjects who improved at least 1 grade in both Evaluator-Reported Submental Fat Rating Scale (ER-SMFRS) and Subject-Reported Submental Fat Rating Scale (SR-SMFRS) | 12 weeks after the final treatment
  Submental Fat Rating Scale is scored on a 5-point scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Percentage of subjects who improved at least 1 grade of Evaluator-Reported Submental Fat Rating Scale (ER-SMFRS) | 4 and 12 weeks after the final treatment
  Submental Fat Rating Scale is scored on a 5-point scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Percentage of subjects who improved at least 1 grade of Subject-Reported Submental Fat Rating Scale (SR-SMFRS) | 4 and 12 weeks after the final treatment
  Submental Fat Rating Scale is scored on a 5-point scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Volume difference of pre-platysmal submental fat around chin area | 4 weeks after the final treatment
  Volume of pre-platysmal submental fat around chin area was measured using MRI
Volume difference of platysmal submental fat around chin area | 4 weeks after the final treatment
  Volume of platysmal submental fat around chin area was measured using MRI
Percentage of subjects who improved at least 2 grades in both Evaluator-Reported Submental Fat Rating Scale (ER-SMFRS) and Subject-Reported Submental Fat Rating Scale (SR-SMFRS) | 4 and 12 weeks after the final treatment
  Submental Fat Rating Scale is scored on a 5-point scale with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Difference of Subject Self Satisfaction Scale (SSSS) | 4 and 12 weeks after the final treatment
  Subject Self Satisfaction Scale (SSSS) assesses participants' satisfaction with their appearance in association with the face and chin on a 7-point scale from 0 to 6 with 0 = Extremely dissatisfied, 1 = Dissatisfied, 2 = Slightly dissatisfied, 3 = Neither satisfied nor dissatisfied, 4 = Slightly satisfied, 5 = Satisfied and 6 = Extremely satisfied.
Difference of Patient-Reported Submental Fat Impact Scale (PR-SMFIS) score | 4 and 12 weeks after the final treatment
  Patients are asked to rate the visual and emotional impact that the appearance of submental fullness had on their self-perception using 11-point scale range from 0 (no impact) to 10 (extreme impact).
Difference of volume of submental fat around chin area analyzed with 3D | 4 weeks after the final treatment
  Volume of submental fat around chin area is measured using a 3D scanner photograph
Patient Global Impression of Change scale (PGIC) | 4 weeks after the final treatment
  Patient global impression of change scale (PGIC) is to rate patients total improvement or worsening in the appearance since before the first treatment compared to final treatment with 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse.
Difference of Derriford Appearance Scale 24 (DAS24) | 4 weeks after the final treatment
  Difference of Derriford Appearance Scale 24 (DAS24) score is to measure distress and dysfunction to problems of appearance with 24 item scale.
Difference of Body Image Quality Life Inventory (BIQLI) score | 4 weeks after the final treatment
  Body Image Quality Life Inventory (BIQLI) assesses participants' body image using 7 point ranging from -3 (very negative) to +3 (very positive).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No